CLINICAL TRIAL: NCT00272051
Title: A Multicenter Randomized Dble-Blind Placebo Controlled Phase III Study of the Efficacy of Xaliproden in Reducing the Neurotoxicity of the Oxaliplatin and 5-FU/LV Combination in First-Line Treatment of Patients With Metastatic Colorectal Carcinoma(MCRC)
Brief Title: XENOX - Evaluation of the Efficacy of Xaliproden in Reducing the Neurotoxicity of the Oxaliplatin + 5-FU/LV Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EFC4972; SR57746A
Record Dates: First submitted 2006-01-03; First posted 2006-01-04 (Estimated); Last update posted 2006-09-13 (Estimated); Status verified 2006-09

CONDITIONS: Metastases; Colorectal Neoplasms; Colorectal Carcinoma
Keywords: Neurotoxicity syndromes; Paresthesia; Oxaliplatin; Xaliproden
MeSH Terms: conditions — Neoplasm Metastasis; Colorectal Neoplasms; Neurotoxicity Syndromes; Paresthesia | interventions — xaliproden

INTERVENTIONS:
Drug: SR57746A

SUMMARY:
Purpose of the trial is to evaluate the efficacy of Xaliproden in reducing the neurotoxicity of the Oxaliplatin and 5-FU/LV chemotherapy, in patients with metastatic colorectal carcinomaPrimary objectives : Compare the risk of occurence of grade 3-4 peripheral sensory neuropathy relative to the cumulative dose of Oxaliplatin between treatment group and placebo group ; Compare the response rate between treatment group and placebo group.Secondary objectives : neurotoxicity parameters (overall incidence, time and dose to onset, time to recovery, change in the sensory action potentials) ; antitumoral efficacy (progression-free survival, overall survival) ; safety profile.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven adenocarcinoma of the colon or the rectum
* age > 18 years
* WHO performance status : 0,1,2
* Signed written informed consent prior to study entry
* Disease stage : metastatic disease not amenable to potentially curative treatment (eg : inoperable metastatic disease)
* Measurable disease
* No prior chemotherapeutic regimen for metastatic disease ; prior adjuvant chemotherapy allowed (disease free interval from end of adjuvant therapy of at least 6 months)
* Prior radiotherapy permitted, if completed at least 3 weeks before randomization, and if not administered to target lesions identified for the study

Exclusion Criteria:

* Chemotherapeutic agents other than 5-FU/LV or 5-FU/Levamizole as part of adjuvant therapy
* Prior therapy with Oxaliplatin
* History of cardiac toxicities under 5-FU/LV therapy or myocardial infarction within the 6 months before study entry ; Known Dihydropyrimidine Dehydrogenase deficiency
* History of intolerance to appropriate antiemetics
* Concurrent active cancer originating from a primary site other than colon or rectum
* Presence of any symptom suggesting brain metastasis
* Known peripheral neuropathy
* Interstitial pneumonia or extensive and symptomatic fibrosis of the lung
* Allergy to Xaliproden/excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 620
Dates: Start 2002-07; Study Completion 2004-05

PRIMARY OUTCOMES:
Clinical evaluation of peripheral sensory neuropathy using the Oxaliplatin specific scale for dose adjustment : Q2W ; response rate using RECIST criteria : Q8W

SECONDARY OUTCOMES:
Safety : Q2W ; Nerve conduction studies : Baseline + cycle 12 ; Progression Free Survival : Q8W ; Survival

CONTACTS AND LOCATIONS:
Overall Officials: Gérard SAID, MD, Study Chair — Hôpital de Bicêtre - Le Kremlin-Bicêtre - France

REFERENCES:
- [Derived] Liu J, Wang X, Sahin IH, Imanirad I, Felder SI, Kim RD, Xie H. Tumor Response-speed Heterogeneity as a Novel Prognostic Factor in Patients With Metastatic Colorectal Cancer. Am J Clin Oncol. 2023 Feb 1;46(2):50-57. doi: 10.1097/COC.0000000000000972. Epub 2022 Dec 26. PMID 36606664
- [Derived] Abdel-Rahman O. Effect of Body Mass Index on 5-FU-Based Chemotherapy Toxicity and Efficacy Among Patients With Metastatic Colorectal Cancer; A Pooled Analysis of 5 Randomized Trials. Clin Colorectal Cancer. 2019 Dec;18(4):e385-e393. doi: 10.1016/j.clcc.2019.07.005. Epub 2019 Jul 15. PMID 31378656
- [Derived] Abdel-Rahman O. Impact of Sex on Chemotherapy Toxicity and Efficacy Among Patients With Metastatic Colorectal Cancer: Pooled Analysis of 5 Randomized Trials. Clin Colorectal Cancer. 2019 Jun;18(2):110-115.e2. doi: 10.1016/j.clcc.2018.12.006. Epub 2018 Dec 28. PMID 30679026
- See also: Related Info — http://www.sanofi-aventis.com